CLINICAL TRIAL: NCT05130814
Title: Perspective Randomized Study Aimed at Evaluating the Effectiveness of the EmoLED Medical Device in the Treatment of Second and Third Stage Pressure Ulcers
Brief Title: EmoLED Medical Device Treatment of Second and Third Stage Pressure Ulcers
Acronym: RISE_UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emoled (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EmoLED_005
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-10

CONDITIONS: Pressure Sore; Pressure Ulcer; Pressure Ulcers Stage III; Pressure Ulcers Stage II
Keywords: ulcer; pressure ulcer; pressure sore; blue light; wound healing; EmoLED; photobiomodulation; LED
MeSH Terms: conditions — Pressure Ulcer; Ulcer | interventions — polyurethane foam; Therapeutics; Bandages

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The Control Group will follow the standard treatment indicated three times a week for the 4 weeks of observation.
  The standard treatment for 2° and 3° stage PU consists of: cleansing with saline or ringer's lactate, hyaluronic acid gauze plus polyurethane foam every 48 hours or as needed. In addition, zinc cream or hyaluronic acid sodium salt + metallic silver is applied to prevent and/or treat the skin maceration of the surrounding area, and eventual debridement of the lesion, application of topical treatment indicated for that stage of the lesion (as provided by the "Protocol on pressure ulcers' dressing" intended as the "standard of care" of the structure) and subsequent bandage (that generally consists of a polyurethane film -thin hydrocolloid plate or a pressure discharge system made with hydrocolloids and polyurethane foam, known as "pressure relief system"), are planned.
  Interventions: Procedure: cleansing; Combination Product: hyaluronic acid gauze plus polyurethane foam; Drug: zinc cream or hyaluronic acid sodium salt + metallic silver; Procedure: topical treatment; Procedure: bandage
- EmoLED Group (Experimental): The Experimental Group will undergo, in addition to the standard treatment, treatment with Emoled three times a week for 4 consecutive weeks.
  This treatment consists of irradiation with the blue light emitted by the device for one minute on the injured area. If the lesion has a greater extension than the irradiated area, multiple repeated applications will be performed, on adjacent areas, until the entire area is covered.
  The treatment with EmoLED will be carried out in correspondence with the dressing change of the lesion.
  Interventions: Device: blue light photobiomodulation; Procedure: cleansing; Combination Product: hyaluronic acid gauze plus polyurethane foam; Drug: zinc cream or hyaluronic acid sodium salt + metallic silver; Procedure: topical treatment; Procedure: bandage

INTERVENTIONS:
Device: blue light photobiomodulation — 1 minute irradiation of blue light performed with EmoLED device.
  Other Names: EmoLED treatment
  Arms: EmoLED Group
Procedure: cleansing — cleaning of the wound area with saline or ringer's lactate
Combination Product: hyaluronic acid gauze plus polyurethane foam — every 48 hours or as needed
Drug: zinc cream or hyaluronic acid sodium salt + metallic silver — applied to prevent and/or treat the skin maceration of the surrounding area
Procedure: topical treatment — topical treatment indicated for that stage of the lesion
Procedure: bandage — it consists of a polyurethane film -thin hydrocolloid plate or a pressure discharge system made with hydrocolloids and polyurethane foam, known as "pressure relief system"

SUMMARY:
The present clinical study aims to verify the effectiveness and safety of the blue light photobiomodulation therapy with EmoLED medical device in supporting the reparative process of the area of the second and third stage decubitus lesion, comparing this method with the effectiveness of the therapy commonly used in the clinical field.

DETAILED DESCRIPTION:
Pressure ulcers (PU), also known as decubitus sores, are areas of lesion localized to the skin and subcutaneous tissue. The development of decubitus ulcers occurs in institutional and community environments, and more frequently in assisted elderly, debilitated and motionless (e.g. orthopedic patients), in patients with severe acute disease (e.g. hospitalized in intensive care units) and in subjects with neurological deficits (e.g. spinal injuries).

Recognizing the considerable economic, health and social impact of pressure ulcers has led to considerable efforts to reduce their occurrence. Nevertheless, pressure ulcers continue to occur. Although not all pressure ulcers are iatrogenic, most of them can be prevented. Pressure ulcers are one of the most frequent iatrogenic lesions in developed countries.

Inadequate treatment methods, such as leaving vulnerable patients in potentially harmful positions for long periods, or massaging reddened skin areas, often continue to be perpetuated even if it has been proven that they are damaging or ineffective.

Pressure, that is often associated to a limitation in mobility of the patient, for a long time has been considered the most important extrinsic factor in the development of pressure ulcers.

However, recent research, and still ongoing, is revealing that shear forces, friction, and microclimate also play an important role in the etiology of pressure ulcers, and that, also, some significant and complex relationships between all these extrinsic factors exist.

In alert patients, the effects of prolonged pressure usually stimulate frequent light body movements to relieve the load and restore tissue perfusion. Unconscious, sedated, anesthetized or paralyzed patients cannot feel or respond to these stimuli and do not move spontaneously. As a result, skin and soft tissue can be exposed to prolonged and without relief pressure.

PUs are generally more common in anatomical locations that cover a bone prominence. In adults, the most common sites are the sacrum and the heel. Other frequently affected anatomical locations are ischium, ankle, elbow and hip.

Pressure ulcers are often difficult to diagnose, in particular it is easy to confuse them with moisture-caused injuries. A correct diagnosis is essential to determine both prevention and treatment plans.

For a proper management of pressure lesions it is essential to take into account their characteristics (location, color, size, amount of exudate, type of tissue, smell, edges) and to consider the condition of the peri-lesional skin (erythema, edema, hardening, maceration). To describe the state of a pressure ulcer, EPUAP (European Pressure Ulcer Advisory Panel) and NPUAP (National Pressure Ulcer Advisory Panel) recommend to divide pressure injuries stages from 1 to 4:

* Stage 1 - Persistent erythema Intact skin with redness not reversible to acupressure in a localized area, usually above a bone prominence. Stage 1 may indicate a patient at risk.
* Stage 2 - Partial thickness tissue loss Loss of the dermis at partial thickness, which looks like a shallow and open ulcer, with red - pinkish lesion bed, without slough. It may also present as a vesicle, intact or open/broken, serous and/or haematic.
* Stage 3 - Total Thickness Tissue Loss Loss of tissue at total thickness. Subcutaneous fat may be visible, but bones, tendons or muscles are not exposed. There may be slough, which does not hide the depth of tissue loss. It may include undermining wounds and tunneling.
* Stage 4 - Loss of subcutaneous tissue Loss of tissue at total thickness with exposure of bones, tendons or muscles. There may be slough or eschar on some parts of the lesion bed. Undermining wounds and tunneling are often present. Stage 4 injuries can extend to muscle and to support structures.
* Not classifiable lesion Loss of tissue at total thickness, where the base of the ulcer is covered by slough (yellow, brown, grey, green or brown) and/or eschar (brown, brown or black) in the bed of the lesion.

The commercial purpose of this study is to value the clinical efficacy of a battery-powered device that uses blue LEDs.

The study aims to compare the response of an existing standard treatment for second and third stage pressure sores, with a protocol that plans the administration of the EmoLED treatment three times a week for 4 consecutive weeks in addition to the conventional therapy.

The Study has an indicative duration of 12 months with an expected enrollment period of 10 months. The study, however, will continue until the number of patients required by this protocol is reached.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 2° or 3° stage lower limb/ sacrum located pressure ulcers;
* Patients with 2° or 3° stage pressure ulcers with a ≥ 2cm² lesion area;
* Patients with a hospitalization waiting time < 30 day;
* Men and women aged ≥ 50 years;
* Patients with a Braden scale score ≥ 11;

Exclusion Criteria:

* Patients who are participating in other clinical trials with drug or medical device;
* Patients with third stage pressure lesions, on the lower limbs or on the sacrum, with undermining wounds, tunneling or eschar;
* Patients with systemic or superficial infection at the time of recruitment, that need systemic antibiotic therapy;
* Patients with a history of self-harm who can voluntarily alter the course of healing;
* Patients under intravenous therapy with doses of corticosteroids above 40mg/day;
* Patients under immunosuppressant or cytostatic drugs therapy;
* Women who are pregnant or breastfeeding1;
* Patients with neoplasia;
* Patients with pathologies that induce skin photosensitivity;
* Patients with a life expectancy of less than 30 days.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Gasperini, Study Director — Medical Advisor; Claudio Macchi, Principal Investigator — IRCCS Don Carlo Gnocchi
Locations (1):
- IRCCS Don Carlo Gnocchi, Florence, Italy

REFERENCES:
- [Derived] Dollaku H, Dalladonna M, Giuliano M, Rossi M, Barbetti P, Marcolongo MS, Buccione E, Iovino P, Macchi C. Randomized clinical trial of the efficacy of the EmoLED medical device in the treatment of stage 2 and stage 3 pressure ulcers: The RISE_UP study. J Tissue Viability. 2025 Aug;34(3):100895. doi: 10.1016/j.jtv.2025.100895. Epub 2025 Mar 26. PMID 40158347

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: The Control Group will follow the standard treatment indicated three times a week for the 4 weeks of observation.
  The standard treatment for 2° and 3° stage PU consists of: cleansing with saline or ringer's lactate, hyaluronic acid gauze plus polyurethane foam every 48 hours or as needed. In addition, zinc cream or hyaluronic acid sodium salt + metallic silver is applied to prevent and/or treat the skin maceration of the surrounding area, and eventual debridement of the lesion, application of topical treatment indicated for that stage of the lesion (as provided by the "Protocol on pressure ulcers' dressing" intended as the "standard of care" of the structure) and subsequent bandage (that generally consists of a polyurethane film -thin hydrocolloid plate or a pressure discharge system made with hydrocolloids and polyurethane foam, known as "pressure relief system"), are planned.
  cleansing: cleaning of the wound area with saline or ringer's lactate
  hyaluronic acid gauze plus polyurethane foam: every 48 hours or as needed
  zinc cream or hyaluronic acid sodium salt + metallic silver: applied to prevent and/or treat the skin maceration of the surrounding area
  topical treatment: topical treatment indicated for that stage of the lesion
  bandage: it consists of a polyurethane film -thin hydrocolloid plate or a pressure discharge system made with hydrocolloids and polyurethane foam, known as "pressure relief system"
- EmoLED Group: The Experimental Group will undergo, in addition to the standard treatment, treatment with Emoled three times a week for 4 consecutive weeks.
  This treatment consists of irradiation with the blue light emitted by the device for one minute on the injured area. If the lesion has a greater extension than the irradiated area, multiple repeated applications will be performed, on adjacent areas, until the entire area is covered.
  The treatment with EmoLED will be carried out in correspondence with the dressing change of the lesion.
  blue light photobiomodulation: 1 minute irradiation of blue light performed with EmoLED device.
  cleansing: cleaning of the wound area with saline or ringer's lactate
  hyaluronic acid gauze plus polyurethane foam: every 48 hours or as needed
  zinc cream or hyaluronic acid sodium salt + metallic silver: applied to prevent and/or treat the skin maceration of the surrounding area
  topical treatment: topical treatment indicated for that stage of the lesion
  bandage: it consists of a polyurethane film -thin hydrocolloid plate or a pressure discharge system made with hydrocolloids and polyurethane foam, known as "pressure relief system"
Period: Overall Study
Arm/Group | Control Group | EmoLED Group
Started | 24 | 24
Completed | 20 | 20
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | EmoLED Group | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Median (Full Range); unit: years] | 75.5 [50 to 91] | 75 [55 to 89] | 75 [50 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 17 | 16 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage Difference in PUSH Score
Description: Change in the index of the PUSH scale of second and third stage ulcers (reflecting the assessment of the clinical state of the lesions) in the two treatment groups at the end of the 4-week observation period. PUSH (Pressure Ulcer Scale for Healing) score is the sum of three subscales measuring wound size (0 to 10), exudate amount (0 to 3) and tissue type (0 to 4). The sum total ranges from 0 (best outcome) to 17 (worst outcome).The change in PUSH scale scores is determined by comparing the mean value at baseline with the final (4-weeks) mean value of the scores obtained for each arm. The comparison was performed by calculating the percentage reduction of the two values; this means that a positive percentage indicates a reduction in the mean values of the PUSH scale and a consequent improvement of the ulcer.
Time Frame: 4 weeks
Population: Per Protocol Analysis
Measure: Mean (Standard Error); unit: percentage reduction of PUSH score
Arm/Group | Control Group | EmoLED Group
Number analyzed (Participants) | 20 | 20
percentage reduction of PUSH score | 23.1 (16.5) | 39.1 (30.0)

2. Secondary Outcome: Change of the Lesion Area
Description: The assessment, during the weeks of observation, of change of the lesion area compared to V0 in the second and third stage lesions in both arms, measured as % of the initial size.The change in ulcer areas is determined by comparing the mean value at baseline with the final (4-week) mean value of areas calculated for each arm. The comparison was performed by calculating the percentage reduction of the two values; this means that a positive percentage indicates a reduction in the mean values of the lesion areas and a consequent improvement of the ulcer.
Time Frame: 4 weeks
Population: Patients with good quality lesion images for image analysis
Measure: Mean (Standard Error); unit: percentage of reduction
Arm/Group | Control Group | EmoLED Group
Number analyzed (Participants) | 13 | 15
percentage of reduction | 29.8 (27.3) | 52.5 (15.6)

3. Secondary Outcome: Number of Treatment-Emergent Adverse Events
Description: Safety of treatment (number of related adverse events in the two groups). All incidents according to the definition of the EU regulation 2017/745 on Medical Devices will be properly reported their gravity and relation with the therapy evaluated.
  It will be counted the number and gravity of occurred adverse events on both arms
Time Frame: 4 weeks
Measure: Number; unit: Number of adverse events
Arm/Group | Control Group | EmoLED Group
Number analyzed (Participants) | 24 | 24
Number of adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of enrollment to the last visit under the protocol (4 weeks, or less in case of healing)
Arm/Group | Control Group | EmoLED Group
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=24) | EmoLED Group (N=24)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT05130814/Prot_SAP_000.pdf